CLINICAL TRIAL: NCT01821586
Title: Optimisation of Oral Rehydration Solution and Evaluation of the Efficacy of Benefiber(Partially Hydrolyzed Guar Gum) Containing Modified Oral Rehydration Solution in the Treatment of Severely Malnourished Children With Watery Diarrhoea
Brief Title: Modified ORS Solution for Severely Malnourished Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-005
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2006-01

CONDITIONS: Malnourished Children With Watery Diarrhoea
Keywords: Diarrhoea;; Severe malnutrition;; Benefiber;; ReSoMal;; modified ORS
MeSH Terms: conditions — Diarrhea; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Modified ORS-1 (Experimental): Modified ORS -1 will be assigned to the enrolled particfipants according to the randomization schedule.
  Interventions: Other: Modified ORS-1
- Modified ORS-2 (ReSoMal) (Experimental): Modified ORS -2 (ReSoMal) will be assigned to the enrolled particfipants according to the randomization schedule.
  Interventions: Other: Modified ORS-2 (ReSoMal)
- Modified ORS-3 (Benefibre) (Experimental): Modified ORS -3 (Benefibre) will be assigned to the enrolled particfipants according to the randomization schedule.
  Interventions: Other: Modified ORS-3 (Benefibre)

INTERVENTIONS:
Other: Modified ORS-1
  Arms: Modified ORS-1
Other: Modified ORS-2 (ReSoMal)
  Arms: Modified ORS-2 (ReSoMal)
Other: Modified ORS-3 (Benefibre)
  Arms: Modified ORS-3 (Benefibre)

SUMMARY:
Diarrhoea and malnutrition are the common childhood illnesses responsible for higher deaths in developing counties. Physiologically, malnourished children excrete lower amounts of salts and water in diarrhoeal stools, and they also are unable to handle excessive salts and water load. Some times they are found to be hyponatraemic due to the shift of sodium inside the cells (inefficient Na+ /K+ pump), and fluids containing higher amounts of sodium (such as the standard ORS) may lead to further increase in the intracellular sodium, fluid overload and heart failure. They also have depleted in potassium stores in the body. Recently, the WHO recommended a special ORS formulation, known as ReSoMal, for management of diarrhoea in severely malnourished children that contains a lower amount of sodium (45mmol/L) and higher amount of potassium (40 mmol/L) than the standard WHO-ORS. It is felt that an ORS containing lower sodium and higher potassium concentration may be useful in correcting hypokalemia, and in lowering the risks of excess sodium and /or overhydration, in severely malnourished children with diarrhoea. The safety of ReSoMaL is, however, still in question due to the risk of hyponatraemia, including symptomatic hyponatraemia, especially in the treatment of severe watery diarrhoea due to Vibrio cholerae and ETEC where loss of sodium in the stool exceeds than that is contained in ReSoMal. Thus an ORS solution with modest concentration of sodium (75 mmol/L) and higher concentration of potassium (40 mmol/L) have been suggested for the treatment of diarrhoea in these children. To improve the efficacy of oral rehydration, in terms of reducing the severity of purging and diarrhoea duration, different approaches (changing the substrates/ reducing the sodium and glucose concentration and osmolarity) have been tried with limited success. Benefiber (partially hydrolysed guar gum), a soluble fiber if added to a ORS solution is expected to be fermented in the colon liberating short chain fatty acids (SCFAs). SCFAs stimulate sodium and water absorption from the colon, and they have trophic effect, act as a fuel source for the colonocytes, have antibacterial properties and stimulates the production commensal flora, thereby may enhance recovery from acute diarrhoea in severely malnourished children. The aims of our proposed study are to examine whether an ORS solution with a modest concentration of sodium will prevent the occurrence of hyponatraemia including symptomatic hyponatraemia, and also whether addition of benefiber will improve the efficacy of ORS solution. This will be a randomized, double blind, controlled clinical trial in 186 children with severe malnutrition and watery diarrhoea (62 in each of the three treatment groups) to compare the efficacy of (i) the currently recommended ORS with some modofication(Na+ 75 mmol/L and K40 momol/L and minerals-Zinc, copper and magnesium), (ii) ReSoMal (Na+ 45 mmol/L), (iii) Currently recommended ORS (Na+ 75 mmol/L, K 40 momol/L and added minerals) with added Benefiber (25 grams/L), in the treatment of acute watery diarrhoea in children with severe malnutrition

DETAILED DESCRIPTION:
Study Design This will be a randomized, double-blind, controlled clinical trial to assess the efficacy of three different modified ORSs: (i) Currently recommended ORS with some modification (Na+ 75, K 40 mmol/L and added minerals); (ii) Resomal (Na+ 45); (iii) Currently recommended ORS (Na+ 75 , K 40 mmol/L and added minerals) with added benefiber (25 grams/L) in the treatment of acute watery diarrhoea in children with severe malnutrition.

STUDY POPULATION Children of either sex, aged 6 months to 3 years, presenting with acute watery diarrhoea of <7 days duration will be screened.

Sample Size

The sample size of this study has been determined based on the followings:

1. Persistence of hyponatraemia: We anticipate that 10% of the children will remain hyponatraemic in the Modified ORS-1 treatment group compared to 30% children in the Modified ORS-2 (ReSoMal). Assuming 5% level of significance and 80% power, the sample size in each group is 60.
2. Recovery from diarrhoea: In a recent clinical trial33 of ORS solution in severely malnourished children with acute watery diarrhoea, the mean +SD duration of diarrhoea was 66 (32) h. We anticipate that a 25% reduction in the diarrhoea duration in children receiving Benefiber-added ORS. Considering 5% level of significance and 80% power the required sample size in each group is 59.
3. Anticipating a drop out of around 5% we need 62 children in each group. Randomization

   After enrolment into the study the patient will be randomized to receive one of the following three solutions:
4. Case Management:

   Following the standardized protocol for management of severely malnourished children used at ICDDR,B hospital 20,23.

   5.1 Fluid therapy (oral) Dehydration will be assessed according to the WHO guidelines, modified for in our last multicentre clinical trial of reduced osmolarity ORS in adult cholera and children with watery diarrhoea (17). In children with some dehydration, the fluid deficit will be corrected with the assigned ORS @ 10ml/kg/hr for the first two hours, then 5ml /kg/hr until the deficit will be corrected. In addition, on going stool looses will be replaced @ 5-10 ml/kg/hr after each watery stool. For high purging patient, the ORS intake will be adjusted according to the ongoing stool loss. ORS therapy will be continued until diarrhoea ceased. Children with severe dehydration, initial rehydration will be done with IV fluid(cholera saline) until the patient is out of shock or disappearance of signs of severe dehydration then the rest of the rehydration will be done as for rehydration in patients with some dehydration as described above.

   5.2 Management of infection: Children without apparent extraintestinal infection will receive Inj ampicillin 100 mg/kg.24 h in 3 divided doses and Inj. Gentamicin @ 5ml/kg.24 h in 2 divided doses for 5 days. Children with lower respiratory tract infection will receive Inj. Ceftriaxone 75 mg /kg.day for 5 days, and those with cholera will receive syrup Azithromycin 20 mg/kg once within 20 minutes of randomization.

   5.3 Diet: Mothers will be advised to continue breastfeeding. Supplementary feeding with milk suji (milk, rice powder mixture, energy 70 kcal/100ml) will be given 10 ml/Kg.feed two hourly for day 1 and increased slowly up to 150 Kcal/Kg.day over 7 days according to demand. If the child has poor appetite, or is weak, or has painful stomatitis or glossitis, food will be delivered through nasogastric tube until able to take food orally. Additionally, semisolid foods (Rice, lentil, vegetable etc.) will be given to older children during convalescent and rehabilitation phase.

   5.4 Vitamin and Mineral Supplements Children older than one year without xeropthalmia will be given 200,000 units of vitamin A and those 6-12 months age will be given 100,000 units of vitamin A on admission. Children with xeropthalmia will receive the same dose on three occasions: on admission, on the following day, and at discharge. Folic acid 1.25 mg and elemental zinc 2 mg/kg will be given until discharge and some medicine will be supplied with the patient to continue upto 15 days. Children will also receive multivitamin drops (1 ml contains Vit A palmitate 5000 IU, vitamin D 1000 IU, thiamine hydrochloride 1.6 mg, riboflavin 1 mg, pyridoxine hydrochloride 1 mg, nicotinamide 10 mg, calcium D- pantothenate 5 mg, and ascorbic acid 50 mg) in a dose of 1 ml twice daily until discharge and some medicine will be supplied with the patient to continue upto 15 days (half the dose for infants, aged <1 year). Hypoglycemia (blood glucose <3.0 mmol/L) will be managed with 50 ml 10% glucose orally or by nasogastric tube. Inj 25% glucose 2 ml/kg will be given if the level of blood glucose below 1.5 mmol/L. Hyponatraemia (serum sodium <115 mmol/L with or without symptoms) will be managed with Inj. 3% NaCl 12 ml/kg I/V slowly over 4 hours.
5. Measurements 6.1 Fluids intakes ( IV, ORS and water) every 6 hours IV fluid will be infused through a calibrated soluset, the amount infused will be noted every 6 hours if the patient is receiving; ORS will be supplied after measuring with a calibrated cylinder and the amount of intake will be noted every 6 hours, if any left over that will be deducted from previous offer. Water will also be measured in a similar way.

6.2 Output (stool, urine and vomit) every 6 hours. Stool will be collected in a bucket of known weight beneath the cholera cot with a central hole and measured every 6 hours with an electronic scale of a precision of 1g. Urine will be collected by pediatric urine collector bag and measured with a calibrated cylinder in ml. Vomit will be collected in a pre-weighed bowl and measured with an electronic scale 6.3 Food intake every 6 hours The children will be offered a defined food of known calorie after measuring with an electronic scale of precision of 1g. Any left over will be measured and subtracted from the amount offered and amount ingested will be recorded every 6 hours. The calorie intake will be estimated from the amount of diet the child consumed.

6.4 Nude body weight will be measured at admission, after rehydration and every 6 hours until recovery of diarrhoea and then at the end of every 24 hours and at discharge

ELIGIBILITY:
Inclusion Criteria:

* Some or severe dehydration (assessed by WHO Guidelines).
* Weight for height (W/H) <70% of NCHS median or with bipedal edema.
* Written informed consent from parents/ guardians

Exclusion Criteria:

* Blood or mucus in stools
* Have received antidiarhoeal drugs for their diarrhoea
* Severe diseases (e.g. severe pneumonia with respiratory distress, clinical sepsis, meningitis) requiring intensive care and other ancillary support like O2 inhalation, oropharyngeal suction etc.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Stool weight | up to 72 hours
  Collection of stool in cholera cot and measured every 6 hours with a using a electronic scale

SECONDARY OUTCOMES:
Duration of Diarrhoea | up to 72 hours
  Time from the onset of randomization upto the stopage of diarrhoea

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Hospital, icddr,b, Dhaka, Bangladesh

REFERENCES:
- [Derived] Alam NH, Ashraf H, Kamruzzaman M, Ahmed T, Islam S, Olesen MK, Gyr N, Meier R. Efficacy of partially hydrolyzed guar gum (PHGG) supplemented modified oral rehydration solution in the treatment of severely malnourished children with watery diarrhoea: a randomised double-blind controlled trial. J Health Popul Nutr. 2015 May 1;34:3. doi: 10.1186/s41043-015-0003-3. PMID 26825757